CLINICAL TRIAL: NCT05076474
Title: An Randomized, Three-treatment, Three-period, Three-sequence, Multiple Dose, Crossover, Comparative Pharmacodynamic Equivalence Study Of Orlistat Capsules 60 mg In Normal, Healthy, Adult, Human Subjects Under Fed Conditions
Brief Title: Pharmacodynamic Equivalence Study Of Orlistat Capsules 60 mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NTP-SEJ-C-BE01
Record Dates: First submitted 2021-09-18; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Orlistat; Capsules

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TR1R2 (Experimental): T(Orlistat 60-mg) R1(Alli 60-mg) R2（Alli 60-mg×2）
  Interventions: Drug: Orlistat 60mg Cap
- R2TR1 (Experimental): R2（Alli 60-mg×2） T(Orlistat 60-mg) R1(Alli 60-mg)
  Interventions: Drug: Orlistat 60mg Cap
- R1R2T (Experimental): R1(Alli 60-mg) R2（Alli 60-mg×2） T(Orlistat 60-mg)
  Interventions: Drug: Orlistat 60mg Cap

INTERVENTIONS:
Drug: Orlistat 60mg Cap — Subjects completed a 5-day run-in period (baseline) and then were randomized to receive the first of 3 treatments; each treatment period lasted 10 days followed by a 4-day washout period between treatments.
  Other Names: Alli Orlistat 60mg Cap; Alli Orlistat 120mg Cap

SUMMARY:
The study will start with a run-in period with controlled diet and no drug for 5 consecutive days. This is to accustom the subjects to the standardized diet and also to determine baseline fecal fat excretion.

After run-in period, subjects will be randomized to receive either test or reference orlistat formulations (60 mg or 120 mg) thrice daily under fed conditions for 10 consecutive days.

DETAILED DESCRIPTION:
To assess the pharmacodynamic equivalence of orlistat, using fat excreted in feces, from sponsor's test product relative to that of reference product in normal, healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* a) Non-smoker, normal, healthy, adult human volunteers with regular bowel movement daily between 18 and 40 years of age (both inclusive).

  b) Having a Body Mass Index (BMI) between 19.0 and 26.0 (both inclusive), calculated as weight in kg/height in m2 and body weight ≥ 50 kg.

  c) Not having significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12 lead ECG, and chest X-ray recordings (P/A view).

  d) Able to understand and comply with the study procedures, in the opinion of the investigator.

  e) Able to give voluntary written informed consent for participation in the trial.

  f) Subjects willing to stay In house for the entire study duration. g) In case of female subjects: Surgically sterilized at least 6 months prior to study participation, Or If of childbearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And Serum pregnancy test must be negative.

Exclusion Criteria:

* a) Known hypersensitivity to orlistat or to any of the excipients of drug. b) History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.

  c) Ingestion of a medicine (including vitamin preparation, herbal remedies, OTC or prescriptions) at any time within 14 days prior to first day of run-in period. In any such case subject selection will be at the discretion of the Principal Investigator.

  d) Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.

  e) Consumption of Grapefruits or grapefruit products within a period of 72 hours prior to receiving the study drug of period-I.

  f) A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc.) or Consumption of alcohol or alcoholic products within 48 hours prior to first day of run-in period.

  g) Smokers, or who have smoked within last six months prior to start of the study.

  h) Difficulty in swallowing solids dosage forms like tablets or capsules. i) The presence of clinically significant abnormal laboratory values during screening.

  j) Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.

  k) History or presence of psychiatric disorders. l) A history of difficulty with donating blood. m) Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.

  n) Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.

  ** If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.

  o) A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.

  p) A positive test result for HIV antibody (1 &/or 2). q) An unusual diet, for whatever reason (for example, fasting, high potassium or low-sodium), for four weeks prior to first day of run-in period. In any such case subject selection will be at the discretion of the Principal Investigator.

  r) Nursing mothers (for female subjects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Fecal fat excretion over 24 hours | 3days
  FFE24= 24h fecal fat content (g)/daily fat (g) *100%

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, Doctor, Principal Investigator — Changsha Third Hospital
Locations (1):
- Shaohong Yin, Linyi, Shandong, China